CLINICAL TRIAL: NCT02289846
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase 2a Study of Oral IW-9179 Administered Once and Twice Daily for 4 Weeks to Patients With Diabetic Gastroparesis
Brief Title: Trial of IW-9179 in Patients With Diabetic Gastroparesis (DGP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-112-202
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo BID (Placebo Comparator): Placebo once in the morning and once in the evening.
  Interventions: Drug: Matching Placebo
- IW-9179 QD AM + Placebo QD PM (Experimental): IW-9179 once in the morning and placebo once in the evening.
  Interventions: Drug: IW-9179; Drug: Matching Placebo
- Placebo QD AM + IW-9179 QD PM (Experimental): Placebo once in the morning and IW-9179 once in the evening.
  Interventions: Drug: IW-9179; Drug: Matching Placebo
- IW-9179 BID (Experimental): IW-9179 once in the morning and once in the evening
  Interventions: Drug: IW-9179

INTERVENTIONS:
Drug: IW-9179
  Arms: IW-9179 BID; IW-9179 QD AM + Placebo QD PM; Placebo QD AM + IW-9179 QD PM
Drug: Matching Placebo
  Arms: IW-9179 QD AM + Placebo QD PM; Placebo BID; Placebo QD AM + IW-9179 QD PM

SUMMARY:
The objectives of this study are to evaluate the safety of IW-9179 in patients with diabetic gastroparesis (DGP) and the effect of treatment on the cardinal symptoms of DGP.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or non-pregnant, non-breastfeeding female, and is age 18 years or older at the time of the Screening Visit.
* Patient has a confirmed diagnosis of type 1 or type 2 diabetes mellitus.
* Patient has a diagnosis of DGP with no history or evidence of mechanical obstruction, symptoms for at least 3 consecutive months preceding the Screening Visit, and delayed gastric emptying of solids documented within 2 years of the Screening Visit.
* Patient has a normal EGD either during the Screening Period or within 2 years of the Screening Visit, with no evidence of structural or organic disease that may explain the patient's gastroduodenal symptoms.
* Patient is compliant with eDiary completion.
* Patient agrees to refrain from making any new, major lifestyle changes.
* Patient is fluent and literate in English.

Exclusion Criteria:

* Patient has a history or current symptoms of any organic or structural disease that, in the opinion of the investigator, can cause abdominal pain or discomfort and may confound the assessment of DGP symptoms.
* Patients with rumination syndrome, cyclic vomiting syndrome, anorexia nervosa, or bulimia.
* Patient is currently using a gastric electric stimulator or has had endoscopic pyloric injections of botulinum toxin within the 6 months prior to the Screening Visit.
* Patient has been hospitalized within the 2 months prior to the Screening Visit for uncontrolled diabetes mellitus, DGP, or associated malnutrition.
* Patient reports significant diarrhea during the four weeks prior to the Screening Visit, or more than 2 days during either week of the Pretreatment Period.
* Patient has had surgery of the GI tract any time before the Screening Visit, an appendectomy or cholecystectomy during the 3 months before the Screening Visit, non-GI surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months, or other major non-GI surgery during the 30 days before the Screening Visit.
* Patient has a history of cancer (resected basal cell or squamous cell carcinoma of the skin is acceptable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Exploratory Endpoint - Daily Severity of Patient-reported Diabetic Gastroparesis Symptoms | Change from baseline: Treatment Period (weeks 1-4) compared with 2-week (baseline) Pretreatment Period

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Ironwood Investigational Site, Birmingham, Alabama
  - Ironwood Investigational Site, Dothan, Alabama
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, North Little Rock, Arkansas
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Los Angeles, California
  - Ironwood Investigational Site, Ventura, California
  - Ironwood Investigational Site, Miami, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, Urbana, Illinois
  - Ironwood Investigational Site, Bastrop, Louisiana
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Rochester, Minnesota
  - Ironwood Investigational Site, Great Neck, New York
  - Ironwood Investigational Site, New York, New York
  - Ironwood Investigational Site, Poughkeepsie, New York
  - Ironwood Investigational Site, Greensboro, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, Webster, Texas
  - Ironwood Investigational Site, Ogden, Utah

REFERENCES:
- [Derived] Ervin CM, Reasner DS, Hanlon JT, Fehnel SE. Exploring the Diabetic Gastroparesis Patient Experience: Patient Exit Interviews. Adv Ther. 2017 Dec;34(12):2680-2692. doi: 10.1007/s12325-017-0632-6. Epub 2017 Oct 27. PMID 29079987